CLINICAL TRIAL: NCT04959422
Title: Assuring Ophthalmologic Follow up for Children Referred Following Instrument-based Vision Screening in a Pediatric Clinic: Effect of Immediate Referral Scheduling and Tracking
Brief Title: Assuring Ophthalmologic Follow up
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled in the study, and staff has been reduced and cannot support the trial any longer.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Andrew J. Schuman, Principal Investigator, Physician, Pediatrics, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02000101
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Vision Screening; Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active scheduling (Experimental): Children who fail instrument vision screens will be scheduled at a community vision specialist office before departure from clinic and all no shows at the vision specialist office will be tracked and rescheduled.
  Interventions: Other: Active scheduling

INTERVENTIONS:
Other: Active scheduling — Active scheduling, tracking and rescheduling, if necessary.

SUMMARY:
The goal of this study is to quantify the improvement in completed ophthalmology referrals and quantify the number of children identified and treated for amblyopia or pre amblyopic strabismus resulting from the implementation of a new referral and tracking system.

DETAILED DESCRIPTION:
Children who fail instrument vision screens at Dartmouth Hitchcock (D-H) Community Group Practice (CGP) Pediatric Clinics will be scheduled at a community vision specialist office before departure from the Pediatric clinic. If the patient does not attend the appointment (a no show) at the vision specialist office , this will be tracked and the patient will be rescheduled.

ELIGIBILITY:
Inclusion Criteria:

* All pediatrics patients without pre-existing vision problems undergoing instrument vision screening at DH Pediatric CGP Clinics in at ages 2,3,4,5, and 6 years of age.

Exclusion Criteria:

* All pediatric patients with pre-existing eye problems that would cause them to be excluded from the study.
* All patients of parents who choose to go to an eyecare provider other than the one participating in the study (as we would be unable to make appointments or track appointments).
* All patients of parents who refuse to make an appointment

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of children who complete vision evaluation | Approximately 1 year
  Number of children who complete vision evaluation with vision specialist

SECONDARY OUTCOMES:
Number of children with amblyopia or pre amblyopic strabismus identified and treated | Approximately 1 year
  Number of children with amblyopia or pre amblyopic strabismus identified and treated with a vision specialist.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Schuman, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Darmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
There are no plan to share IPD at this time.